CLINICAL TRIAL: NCT00100373
Title: Characterization of the Immune Response and Viral Shedding to Experimental Infection With Respiratory Syncytial Virus, Strain A-2, in Healthy Adults Ages 21 to 40 Years Old
Brief Title: RSV Challenge in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 04-035
Record Dates: First submitted 2004-12-30; First posted 2004-12-31 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2007-02

CONDITIONS: Respiratory Infections, Acute; Respiratory Syncytial Virus
Keywords: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Tract Infections; Respiratory Syncytial Virus Infections

INTERVENTIONS:
Drug: RSV challenge material

SUMMARY:
The purpose of this study is to measure the immune response (how the body fights infection) to an experimental preparation of live Respiratory Syncytial Virus (RSV). A better understanding of this virus may be useful in development of vaccines and treatments. Participants will include 20 healthy adults age 21-40. Study procedures will include drawing blood, urine samples, respiratory exams, vital signs and temperature, diary cards, nasal mucus weight and nasal washes and swabs. All participants will receive vaccine via nose drops. Patients will participate in the study for about 2 months.

DETAILED DESCRIPTION:
Respiratory infections are a major cause of morbidity and mortality in the elderly. Recently, respiratory syncytial virus (RSV) has been shown to account for a significant portion of these illnesses. The causative factors associated with severe RSV disease in the elderly are not well understood. The contribution of viral load, host inflammatory responses and the cellular immune response to disease pathogenesis are unknown. A better understanding of these processes may be useful in the development of vaccines and therapeutics for RSV disease. Although the adult groups at highest risk for serious RSV disease are elderly and high-risk adults, we propose to use the challenge model in young healthy adults to determine optimal timing of specimen collection and the feasibility of performing certain tests before moving ahead to the target groups with natural infection. The purpose of this study is to measure the immune response (how the body fights infection) to an experimental preparation of live Respiratory Syncytial Virus (RSV. Participants will include 20 healthy adults age 21-40. Study procedures will include drawing blood, urine samples, respiratory exams, vital signs and temperature, diary cards, nasal mucus weight and nasal washes and swabs. All participants will receive vaccine via nose drops. Patients will participate in the study for about 2 months.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults ages 21 to 40 years. Able to and has given informed consent to participate. Negative urine pregnancy test, if female. Pre-challenge serum neutralizing titer to RSV A2 by microneutalization (MNA) of </= 1:657 (9.36 log2) Non-smoker No significant health abnormalities detected by evaluation of medical history, general physical examination, vital signs and laboratory tests.

Willingness to remain in isolation for 11 nights and comply with all study requirements.

Willingness to remain in the Rochester area for the 28 days of the study.

Exclusion Criteria:

Volunteers with any of the following conditions will not be eligible to participate:

Chronic medical conditions requiring medical followup within the last 6 months. Serologic evidence of infection with HIV or hepatitis C virus, or presence of hepatitis B surface antigen in serum.

History of medically documented asthma requiring treatment (including over-the-counter medications) at any time.

Any abnormal laboratory results which would render challenge with RSV unsafe or interfere with the interpretation of the subject's response to challenge, e.g., AST, ALT, Bilirubin, BUN, creatinine. ( see Appendix II) Individuals requiring concurrent therapy with medications likely to interfere with evaluation of the response to infection, e.g. antipyretics, anti-inflammatory medications Close contact with children aged less than 2 years, with any individuals with significant immunosuppression, or with individuals greater than 65 years of age.

Health care workers with any patient contact during the two weeks following challenge Pregnancy or uncertain status regarding pregnancy Acute respiratory infection or fever within 1 week of challenge Previous enrollment in a study evaluating RSV challenge viruses or RSV vaccines.

Known glucose intolerance (history of abnormal glucose tolerance test or medical history of diabetes mellitus).

History of chronic obstructive disease, emphysema or other serious or evolving pulmonary disease.

Any condition in the opinion of the investigator might interfere with study objectives or pose excessive risks to subjects.

History of previous hospitalization for a pulmonary condition (ie. Pneumonia, asthma, spontaneous pneumothorax, or severe sinus disease requiring a surgical procedure.

History of frequent serious bacterial infections associated with low white blood cell count (below 4,000 per microgram)

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13
Dates: Start 2004-09; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Locations (1):
- Rochester General Hospital, Rochester, New York, United States